CLINICAL TRIAL: NCT02181556
Title: Efficacy and Safety of Aflibercept in Combination With FOLFIRI Chemotherapy as 1st Line Treatment for Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FFCD 1302
Record Dates: First submitted 2014-07-02; First posted 2014-07-04 (Estimated); Results first posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-05

CONDITIONS: Metastatic Colorectal Cancer
Keywords: colorectal cancer; Metastatic
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — IFL protocol; aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FOLFIRI + Aflibercept (Experimental): FOLFIRI and aflibercept (4 mg/m²) each 14 days until progression of disease
  Interventions: Drug: FOLFIRI Protocol; Drug: Aflibercept Injection

INTERVENTIONS:
Drug: FOLFIRI Protocol — injection of FOLFIRI and Aflibercept every 14 days until progression of disease
Drug: Aflibercept Injection — injection of FOLFIRI and Aflibercept every 14 days until progression of disease

SUMMARY:
One of the treatments generally used to treat this disease is a chemotherapy called FOLFIRI. The purpose of this study is to improve the efficacy of the chemotherapy by adding a protein, similar to immunoglobulins, aflibercept, and to assess their tolerance.

Aflibercept is a protein that has already been studied in the treatment of metastatic colorectal cancers, in combination with a chemotherapy involving irinotecan in addition to 5FU (fluoropyrimidine) ( (FOLFIRI) as 2nd line treatment. It is marketed in Europe and it is authorized in the United States. Its addition to this chemotherapy combination has in fact brought about a benefit in terms of progression-free survival and overall survival.

The purpose of the study is to evaluate the efficacy and tolerance of this combination rather in the initial approach to the treatment of metastatic colorectal cancers and hence to evaluate it as 1st line treatment

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Overall state as per WHO (World Health Organization) ≤ 2
* Life expectancy > 3 months
* Metastatic adenocarcinoma of the rectum or of the colon histologically proven on the primary tumor or a metastasis
* Unresectable metastasis (metastases) and/or inoperable patient
* Patient eligible for a 1st line treatment associating 5 FU-Irinotecan (FOLFIRI) and aflibercept
* At least one measurable target lesion according to RECIST criteria v1.1 not previously irradiated
* Absence of prior treatment of the metastatic disease. Prior adjuvant chemotherapy completed at least 12 months before the metastatic cancer diagnosis is authorized
* Satisfactory laboratory panel: Hb> 9 g/dl, polynuclear neutrophils > 1500 /mm3, platelets > 100,000/mm3, total bilirubin < 1.5 x UNL(upper normal limit), creatinine clearance > 50 mL/min (cockcroft-Gault formula - appendix 4), PAL (alkaline phosphatase) < 5 x UNL, AST (aspartate aminotransferase) and ALT (alanine aminotransferases) < 5 x UNL, GGT (gamma-glutamyltransferase) < 5 x UNL,
* Proteinuria on urine dipstick < 2+. If > 2+ test 24-hour proteinuria, which should be < 1 g

Exclusion Criteria:

* Patients whose primary tumor is in place and presenting clinical symptoms (occlusion; hemorrhage)
* Brain metastases
* Gilbert's syndrome
* Uncontrolled hypercalcemia
* Hypertension not kept under control (SBP (Systolic Blood Pressure) >150 mmHg and DBP (Diastolic Blood Pressure) >100 mmHg) or history of hypertensive crisis or hypertensive encephalopathy
* Any unbalanced active disease over the last 6 months: liver failure, kidney failure, respiratory failure, congestive heart failure, unstable angina, myocardial infarction, significant arrhythmia (Patients treated by anticoagulants (coumadin, warfarin) are eligible if strict monitoring of the INR( international normalized ratio) is possible)
* Significant surgical intervention within the 28 days before the start of treatment
* Presence of active gastroduodenal ulcer, non-healed wound or bone fracture
* Antitumor treatments other than those included in the study (chemotherapy, targeted therapy, immunotherapy)
* History of malignant hemopathy or cancer except for those treated more than 5 years ago and considered healed, in situ carcinomas of the uterine cervix and treated skin cancers (except for melanoma)
* Pregnant or breast-feeding women, women of childbearing age not having taken a pregnancy test, absence of effective contraception in patients (men and/or women) of childbearing age
* Any contraindication of the drugs used in the study
* Impossible to meet the medical follow-up requirements of the study for geographic, social or psychological reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julien TAIEB, PhD, Principal Investigator — Fédération Francophone de Cancérologie Digestive
Locations (8):
- France (8):
  - CHU - Hôtel Dieu, Angers
  - Hôpital Avicenne, Bobigny
  - CHU - Hôpital François Mitterand, Dijon
  - Clinique Jean Mermoz, Lyon
  - La Timone, Marseille
  - Hôpital Européen Geaorge Pompidou (HEGP), Paris
  - Hôpital La Pitié Salpetière, Paris
  - Hôpital Trousseau, Tours

REFERENCES:
- [Result] Lapeyre-Prost A, Pernot S, Sigrand J, Le Malicot K, Mary F, Aparicio T, Dahan L, Caroli-Bosc FX, Lecomte T, Doat S, Marthey L, Desrame J, Lepage C, Taieb J. Aflibercept in Combination With FOLFIRI as First-line Chemotherapy in Patients With Metastatic Colorectal Cancer (mCRC): A Phase II Study (FFCD 1302). Clin Colorectal Cancer. 2020 Dec;19(4):285-290. doi: 10.1016/j.clcc.2020.06.003. Epub 2020 Jun 12. PMID 32921581

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 41 patients were included by 9 centers between October 2014 and February 2017
Period: Overall Study
Arm/Group | FOLFIRI + Aflibercept
Started | 41
Completed | 40
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | FOLFIRI + Aflibercept
Number analyzed (Participants) | 40
Age, Continuous [Median (Full Range); unit: years] | 64.85 [45.72 to 80.39]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 40

OUTCOME MEASURES:

1. Primary Outcome: Rate of Patients Alive and Progression-free 6 Months After Inclusion.
Description: Progression was evaluated by CT scan, according to RECIST criteria (version 1.1) definition by the investigator. Death was also considered as an event (all causes).
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions compared the little sum of diameters observed during the study (NADIR), or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 6 months
Population: Analyse was done on all the patients included in the study (ITT)
Measure: Number; unit: Nb of patients alive without progression
Arm/Group | FOLFIRI + Aflibercept
Number analyzed (Participants) | 40
Nb of patients alive without progression | 22

2. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from the date of the patient's inclusion to the patient's death (all causes). For alive patients the date of the latest news is taken into account
Time Frame: Up to 2 years after the end of the treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | FOLFIRI + Aflibercept
Number analyzed (Participants) | 40
Months | 18.63 [14.69 to 30.65]

3. Secondary Outcome: Progression-free Survival
Description: The progression-free survival is the time from inclusion to the first radiological progression or death (all causes). For patients alive without progression date of last news will be considered.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions compared the little sum of diameters observed durin the study (NADIR), or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: up to 12 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | FOLFIRI + Aflibercept
Number analyzed (Participants) | 40
Months | 8.16 [6.11 to 10.38]

ADVERSE EVENTS:
Time Frame: Up to the end of treatment, on average of 8 months
Description: Toxicities were collected before each cure of treatment up to the end of the treatment. There is no fixed time-frame because of metastatic disease. The study treatment is given until withdrawal of the patients for any reason (Toxicities, progression or any other medical reason)
Groups:
- FOLFIRI and Aflibercept: FOLFIRI and aflibercept (4 mg/m²) each 14 days until progression of disease
  FOLFIRI + Aflibercept: injection of FOLFIRI and Aflibercept every 14 days until progression of disease
Arm/Group | FOLFIRI and Aflibercept
All-Cause Mortality (participants affected / at risk) | 25/40
Serious Adverse Events (participants affected / at risk) | 13/40
Other Adverse Events (participants affected / at risk) | 36/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOLFIRI and Aflibercept (N=40)
Abdominal Pain (Gastrointestinal disorders) | 3 (4)
Anal fistula (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Decreased appetite (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FOLFIRI and Aflibercept (N=40)
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 5
Abdominal Pain (Gastrointestinal disorders) | 5
Mucositis (Gastrointestinal disorders) | 6
Colonic perforation (Gastrointestinal disorders) | 2
Venous TE disorders (Vascular disorders) | 7
Hypertension (Vascular disorders) | 7
Proteinuria (Renal and urinary disorders) | 2
Anemia (Investigations) | 2
Leucopenia (Investigations) | 2
Neutropenia (Investigations) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2014-01-24): https://cdn.clinicaltrials.gov/large-docs/56/NCT02181556/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-14): https://cdn.clinicaltrials.gov/large-docs/56/NCT02181556/SAP_001.pdf